CLINICAL TRIAL: NCT02768402
Title: Percutaneous Mitral Valve Replacement EvaLuation Utilizing IDE Early Feasibility Study (PRELUDE)
Brief Title: Caisson Transcatheter Mitral Valve Replacement (TMVR) System Early Feasibility Study
Acronym: PRELUDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Caisson Interventional LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral Valve Regurgitation; Primary MR; Secondary MR; MR; Heart Failure; Structural Heart; Secondary Mitral Valve Regurgitation; Primary Mitral Valve Regurgitation; Transseptal; Transcatheter
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): All eligible patients will be in the treatment arm for the 'Caisson TMVR System' (transcatheter mitral valve replacement) procedure. No control or comparator in this study.
  Interventions: Device: Caisson TMVR System

INTERVENTIONS:
Device: Caisson TMVR System — Transcatheter mitral valve replacement is a percutaneous procedure used to treat mitral valve regurgitation with a prosthetic valve implantation.

SUMMARY:
The purpose of this study is to assess the safety and performance of the Caisson Interventional Transcatheter MitralValve Replacement (TMVR) system for the treatment of severe symptomatic MitralValve Regurgitation (MR).

DETAILED DESCRIPTION:
The treatment guidelines for valvular heart disease indicate that surgical correction of primary mitral valve regurgitation (MR) is a Class I recommendation. Further, recent evidence indicates that valve replacement is at least as effective as repair in both primary and secondary MR patients. However, many patients are not referred for surgery as they are considered to be too high of a risk to undergo on pump, open-heart procedures. Percutaneous aortic valve replacement has made treatment of stenosed aortic valves available to high-risk surgical patients who would have otherwise been medically managed. Percutaneous mitral valve (MV) replacement offers similar advantages. Currently, the only approved percutaneous treatment for MR is MitraClip. MitraClip is limited to a specific population of high risk surgical patients with valvular prolapses that are amenable to repair by the edge to edge technique. The feasibility of percutaneous MV replacement has been shown in animal studies, the implantation of aortic valves at the mitral position, and early evaluations of purpose made transcatheter MVs in humans. To meet this medical need, Caisson Interventional has developed a percutaneous delivery system for a bioprosthetic mitral valve. As with patients with aortic valve (AV) deficiencies, this device can be used to provide needed therapy to patients who might not otherwise receive treatment beyond medical therapy. This study will provide initial information on the safety and performance of this system.

ELIGIBILITY:
Inclusion Criteria:

* Has severe mitral regurgitation
* New York Heart Association (NYHA) Class II, III, IVa or heart failure
* High risk for cardiovascular surgery

Exclusion Criteria:

* Excessive calcification or thickening of mitral valve annulus, severe mitral stenosis, fused commissures, valvular vegetation or mass
* Left ventricular end diastolic dimension > 7cm
* Left ventricular outflow tract obstruction
* Severe right ventricular dysfunction
* Stroke within 90 days; transischemic attack or myocardial infarction within 30 days of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients without Major Adverse Events (MAEs) | 30 days
  Freedom from major adverse events including death, stroke, myocardial infarction and surgical reintervention through 30 days

SECONDARY OUTCOMES:
Number of patients with successful delivery and implantation of the prosthetic valve (technical success) | Intraoperative
  Successful delivery and retrieval of the transcatheter mitral valve delivery system; deployment and correct positioning (via intraoperative imaging) in the appropriate anatomic location of prosthetic valve with no requirement for additional surgery
Number of living, stroke-free patients with prosthetic valve in place (device success) | 30 days
  Patient is alive, stroke-free, original intended device in place (echo), no mitral valve surgical re-intervention required

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Williams, MD, Study Director — NYU Langone Medical Center
Locations (13):
- United States (13):
  - Cedars Sinai Medical Center, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Delray Medical Center, Delray Beach, Florida
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth, Columbus, Ohio
  - Saint Thomas Heart, Nashville, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Health Services, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No